CLINICAL TRIAL: NCT01184456
Title: A Controlled Trial to Evaluate the Effects of GanedenBC30 on the Immune System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Healthcare Foundation (Other)
Collaborators: Ganeden Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHF-GAN01
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: HIV Infection; Gastrointestinal Symptoms
Keywords: AIDS; Acquired Immunodeficiency Syndrome; HIV; Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — exopolysaccharide biopolymer, Bacillus coagulans; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GanedenBC30, GBI-30, PTA-6086 (Experimental)
  Interventions: Dietary Supplement: GanedenBC30, GBI-30, PTA-6086
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: GanedenBC30, GBI-30, PTA-6086 — 1 capsule per day containing 2 billion CFU of GanedenBC30, GBI-30, PTA-6086 for 90 days.
  Other Names: Bacillus coagulans; Probiotics
  Arms: GanedenBC30, GBI-30, PTA-6086
Drug: Placebo — 1 capsule per day for 90 days.
  Arms: Placebo

SUMMARY:
Improvement in the rate of bacterial translocation may lead to a decrease in a chronic inflammatory response thereby decreasing CD4 destruction and HIV proliferation.

By the addition of probiotics we hope to show a reduction in LPS leading to a decrease in chronic inflammation and therefore an improvement in immune markers.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or non-pregnant, non-lactating female.
* Adults 18 years or older.
* Is able to provide written, informed consent to participate in the study.
* Serological documentation of HIV infection at any time prior to study entry and is clinically stable.
* Stable CD4 count greater than or equal to 250 cells/cubic mm for six months prior to study entry (+/- 50 cells/cubic mm).
* HIV-1 RNA ≤50 copies/mL for six months prior to study entry.
* Karnofsky performance status - 60%.
* Adequate laboratory parameters within the last 30 days:

  1. absolute neutrophil count >1000 cells/cubic mm
  2. hemoglobin >9.0 g/dL
  3. platelets >75,000/cubic mm
  4. creatinine <1.5 x upper limit of normal
  5. SGOT/SGPT <3.0 x upper limit of normal
  6. bilirubin <2.0 mg/dL
* Patients with documented GI symptoms to include but are not limited to: flatulence, diarrhea, bloating, gastroesophageal reflux disease, nausea, and constipation.
* If females are of childbearing potential, they must be practicing an effective method of contraception and agree to use birth control while on protocol and for 1 month after completion of study. Women of Child Bearing Potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to start of study medication. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not. postmenopausal [defined as amenorrhea for 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL]. Even women who are using oral, implanted or, injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential.
* Must agree to practice protected sexual activity (via barrier method) during course of the study.
* In the opinion of the investigator, is willing and able to comply with the study requirements.

Exclusion Criteria:

* Active opportunistic infection, which is progressive, or imminently disabling or life threatening, in the judgment of the Principal Investigator with exception of Kaposi Sarcoma.
* Cytotoxic chemotherapy, interferon treatment, or radiation therapy within the preceding 3 weeks (subjects who have received intralesional chemotherapy will not be excluded, however).
* Any antibiotic therapy within 30 days of enrollment
* Any probiotic formulation within 30 days of enrollment
* Any immunization within 30 days of enrollment
* Known history of allergic reactions to any of the investigational products or their ingredients.
* Chronic treatment with immunosuppressant drugs, including corticosteroids, except for the treatment of adrenal insufficiency. Topical steroids are permitted.
* History of or known current malabsorption syndrome.
* Any grade 3 or 4 lab abnormalities as defined by a standardized grading scheme based on the DAIDS table (see Appendix B) with the following exceptions:
* Pre-existing diabetes with glucose toxicity elevations ≥ grade 3
* Triglyceride or total cholesterol elevations ≥ grade 3
* Clinical or laboratory evidence of clinically significant liver impairment/ dysfunction, disease or cirrhosis.
* Life expectancy < 6 months in the opinion of the investigator.
* Active substance abuse or significant psychiatric illness that in the opinion of the investigator might interfere with study compliance.
* Female subject of childbearing potential not using effective non-hormonal birth control methods or not willing to continue practicing these birth control methods from screening until the last trial related activity.
* Subject is pregnant or lactating.
* Any condition that in the Principal Investigator's opinion may render the subject unable to complete the study or which may pose significant risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AHF Research Center, Beverly Hills, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PI has left AIDS Healthcare Foundation, all efforts to locate the data have been exhausted and no data is available.
Period: Overall Study
Arm/Group | GanedenBC30, GBI-30, PTA-6086 | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: PI has left AIDS Healthcare Foundation, all efforts to locate the data have been exhausted and no data is available.
Groups:
- Total: Total of all reporting groups
Arm/Group | GanedenBC30, GBI-30, PTA-6086 | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Effects of Daily Consumption of GanedenBC30 on Immune Function and Gastro-intestinal Issues
Description: The primary endpoint measurement of safety is measured based on the number of adverse events reported relative to the expected number adverse events prior to the start of the study based on a risk analysis.
  The primary endpoint measurement of immune function is measured based on biological markers including CRP, IL-8 and TNF-alpha between the two groups.
  The primary endpoint measurement of gastro-intestinal issues is measured based on the number of reported symptoms relative to the expected number of gastro-intestinal issues prior to the start of the study based on a risk analysis.
Time Frame: 30, 60, and 90 days.
Population: PI has left AIDS Healthcare Foundation, all efforts to locate the data have been exhausted and no data is available.
Arm/Group | GanedenBC30, GBI-30, PTA-6086 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: PI has left AIDS Healthcare Foundation, all efforts to locate the data have been exhausted and no data is available.
Description: PI has left AIDS Healthcare Foundation, all efforts to locate the data have been exhausted and no data is available.
Arm/Group | GanedenBC30, GBI-30, PTA-6086 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No